CLINICAL TRIAL: NCT05207085
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose Titration Study to Assess the Safety, Tolerability, and Efficacy of Valbenazine for the Treatment of Trichotillomania in Adults
Brief Title: Efficacy of Valbenazine for the Treatment of Trichotillomania in Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000034993; 2000026788 (Other: Yale)
Record Dates: First submitted 2021-12-21; First posted 2022-01-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Trichotillomania (Hair-Pulling Disorder)
Keywords: trichotillomania; hair-pulling disorder; valbenazine
MeSH Terms: conditions — Trichotillomania | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Valbenazine (Experimental): Participants randomized1:1 to receive valbenazine
  Interventions: Drug: Valbenazine Oral Capsule
- Placebo (Placebo Comparator): Participants randomized 1:1 to receive placebo
  Interventions: Other: Placebo Oral capsule

INTERVENTIONS:
Drug: Valbenazine Oral Capsule — Participants randomized to active treatment will be given a starting dose of 40mg of valbenazine , which may be escalated to 80mg to achieve an optimal dose of the medication for each subject.
  Other Names: Ingrezza
  Arms: Valbenazine
Other: Placebo Oral capsule — Participants randomized to placebo will be given a capsule that is the same shape and color as the active medication and will subject to the same dose escalation requirements as the other arm but will receive placebo during the treatment period.
  Arms: Placebo

SUMMARY:
This trial aims to evaluate the efficacy, safety and tolerability of valbenazine, titrated to the subject's optimal dose of 40mg or 80mg, administered once daily, for 12 weeks, for the treatment of trichotillomania (TTM) in a double blind placebo controlled design study. After week 12, subjects will begin a 12-week, open-label portion of the study. During the open-label portion of the study, all subjects will receive the study drug at their optimal dose. The primary endpoint of these studies will be the change from baseline of placebo vs. active scores utilizing the Massachusetts General Hospital Hairpulling Scale (MGH-HPS) at the end of Week 12.

DETAILED DESCRIPTION:
Eligible subjects will be randomized in a double-blind manner in a 1:1 ratio to once-daily doses of valbenazine or placebo for 12 weeks. After week 12, all subjects will begin the 12-week, open-label portion of the study in which they all get their optimal dose. Follow-up assessments will be conducted at the end of week 26 (2 weeks after the last dose of the study drug). For subjects randomized to active treatment, the starting dose will be valbenazine 40mg, which may be escalated to 80mg to achieve an optimal dose of valbenazine for each subject. Dose escalation will occur at the end of week 2 based on the following criteria: 1) the subject's TTM symptoms are not sufficiently controlled per physician investigator assessment and 2) an evaluation by the physician investigator indicates that the subject is tolerating the study drug at the current dose and would likely be able to tolerate the higher dose level. At week 4, the physician investigator may choose to keep the subject at the higher dose or may reduce to the subject's prior tolerated dose (in subjects who have had dose escalation). If a subject's optimal dose was established as 40mg at week 2, no dose escalation will be allowed at week 4. At any time after week 2, the physician investigator may decrease the dose to the previous dose for any subject who had a dose escalation and who is unable to tolerate a given dose increase. The investigator may reduce the subject's dose only one time. Subjects who are unable to tolerate the starting dose or resumption of the 40mg dose will be discontinued from the study. The subject will continue at the dose reached during the optimization period for the remainder of the 12-week treatment period. To maintain the study blind, subjects randomized to placebo in each weight group will be subjected to the same dose escalation requirements, but will receive only placebo during the treatment period. Following the 12-week, double-blind study, all subjects will be offered the option to receive open-label valbenazine for 12 weeks. In order to protect the blind in the first phase of the trial all subjects will receive 40mg of valbenazine from week 12 to week 14 and then be titrated on the study medication similar to the first phase of the trial from that point forward.

ELIGIBILITY:
Inclusion Criteria:

1. Have documentation of written and witnessed consent from the subject.
2. Male or female adult between the ages of 18-65, inclusive.
3. Be in good health as determined by medical history, physical examination, laboratory assessments and 12-lead ECG.
4. On stable psychiatric medication regime of 4 weeks prior to beginning the trial and not anticipating changes during the trial.
5. Subjects of child-bearing potential must agree to use contraception (condoms for men, birth control pill or diaphragm for women) consistently from screening until 30 days (female) or 90 days (male) after the last dose of the study drug. A female subject of childbearing potential is defined as a female capable of becoming pregnant, which includes subjects who have had their first menstrual cycle (i.e., menarche) and are not surgically sterile (i.e., bilateral oophorectomy, hysterectomy or bilateral tubal ligation for at least 3 months prior to screening) or have not experienced menopause and subsequently are no longer of childbearing potential. A male subject of childbearing potential is defined as a subject who has reached spermarche and has not been vasectomized for at least 3 months prior to screening. Subjects who practice total abstinence from sexual intercourse as the preferred lifestyle are not required to use contraception (periodic abstinence is not acceptable).
6. Female subjects must have a negative urine pregnancy test at screening, baseline and weeks 2, 4, 8, 12, 14, 16, 20, 24 and 26.
7. Negative urine drug screen (negative for amphetamines, barbiturates, benzodiazepine, phencyclidine, cocaine, or opiates) at screening, baseline and weeks 2, 4, 8, 12, 14, 16, 20, 24 and 26. Subjects on stable doses of prescribed and supervised (not as needed) benzodiazepines, opiates or psychostimulants (participants with ADHD) can participate in the study. Results from a positive drug screen will be discarded.
8. Be willing to adhere to the study regime and study procedures described in the protocol and informed consent forms, including all requirements at the study center and return for the follow-up visit.
9. Have symptoms that cause marked distress or significant impairment in occupational and/or social function.
10. Have a stable psychiatric status (TTM) as clinically determined by the investigator.
11. Meet DSM-5 criteria for TTM.
12. Significant current TTM symptoms: 12 or greater score on MGH-HPS.

Exclusion Criteria:

1. Comorbid bipolar disorder, psychotic disorder, substance use disorder, developmental disorder or intellectual disability (IQ<70).
2. Recent changes in medications (less than 4 weeks) in other medications that have potential effects on TTM severity. Medication change is defined to include dose changes or medication discontinuation.
3. Currently taking antipsychotic medications or other medications that affect the dopamine system (e.g. psychostimulant medications).
4. Recent changes in behavior treatment (less than 4 weeks) or initiation of therapy (within 12 weeks) for TTM/Obsessive Compulsive Disorder (OCD).
5. Taking co-medications (over the counter or prescription) that may have a drug interaction with valbenazine as described in the United States Prescribing Information for INGREZZA. Patients who are taking co-medications with the potential to cause QT prolongations will not be excluded unless their ECG shows QT prolongation already present.
6. Positive pregnancy test or drug screening test.
7. Currently pregnant or lactating.
8. Significant medical comorbidity.
9. Excessive use of tobacco and/or nicotine-containing products (based on the investigator's assessment or more than 1½ pack of cigarettes per day, 1 can of chewing/dipping tobacco per day, 54mg of nicotine-containing smoking cessation products per day, or any nicotine products or combination of products that exceed 54mg per day) within 30 days of screening.
10. History of substance (drug or alcohol) dependence or abuse within 3 months before Baseline, as defined by DSM-5 criteria for Substance Use Disorder.
11. Known history of neuroleptic malignant syndrome.
12. Known history of long QT syndrome or cardiac arrhythmia.
13. Have a screening or Day 1 average triplicate ECG corrected QT interval using Fridericia's formula (QTcF) of >450msec or the presence of any clinically significant cardiac abnormality.
14. Have a blood loss ≥250 mL or donated blood within 56 days or donated plasma within 7 days of Day 1 (baseline).
15. Have a significant risk of suicidal or violent behavior based on prior medical history and clinical judgement.
16. Have an allergy, hypersensitivity, or intolerance to VMAT2 inhibitors (e.g., tetrabenazine).
17. Have a history of or suspected poor compliance in clinical research studies.
18. Have previous experience with valbenazine or previously participated in a valbenazine clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in Massachusetts General Hospital Hairpulling Scale (MGH-HPS) from baseline to Week 12 | baseline to week12
  Massachusetts General Hospital Hairpulling Scale (MGH-HPS) scores range from 0-28 with 28 being the most severe. The lower the total score, the lower the severity level. This scale is given and measured once every 2 weeks for a total of 12 weeks.

SECONDARY OUTCOMES:
Clinical Global Improvement Scale - Trichotillomania Severity (CGI-TTM) score at endpoint | Week 12
  Each of the Clinical Global Improvement Scale -Trichotillomania (CGI-TTM) response categories was assigned a numerical score as follows: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = Not changed; 5 = Minimally worse; 6 = Much worse; 7 = Very much worse. Responder status on Clinical Global Improvement Scale as having a CGI-TTM score at endpoint less than or equal to 2.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Bloch, MD, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] United States Prescribing Information for INGREZZA. San Diego, CA 92130: Neurocrine Biosciences, Inc.; 2020.
- [Background] Grant JE, Chamberlain SR. Trichotillomania. Am J Psychiatry. 2016 Sep 1;173(9):868-74. doi: 10.1176/appi.ajp.2016.15111432. PMID 27581696
- [Background] Bloch MH, Landeros-Weisenberger A, Dombrowski P, Kelmendi B, Wegner R, Nudel J, Pittenger C, Leckman JF, Coric V. Systematic review: pharmacological and behavioral treatment for trichotillomania. Biol Psychiatry. 2007 Oct 15;62(8):839-46. doi: 10.1016/j.biopsych.2007.05.019. Epub 2007 Aug 28. PMID 17727824
- [Background] McGuire JF, Ung D, Selles RR, Rahman O, Lewin AB, Murphy TK, Storch EA. Treating trichotillomania: a meta-analysis of treatment effects and moderators for behavior therapy and serotonin reuptake inhibitors. J Psychiatr Res. 2014 Nov;58:76-83. doi: 10.1016/j.jpsychires.2014.07.015. Epub 2014 Jul 26. PMID 25108618
- [Background] Franklin ME, Zagrabbe K, Benavides KL. Trichotillomania and its treatment: a review and recommendations. Expert Rev Neurother. 2011 Aug;11(8):1165-74. doi: 10.1586/ern.11.93. PMID 21797657
- [Background] Sarva H, Henchcliffe C. Valbenazine as the first and only approved treatment for adults with tardive dyskinesia. Expert Rev Clin Pharmacol. 2018 Mar;11(3):209-217. doi: 10.1080/17512433.2018.1429264. Epub 2018 Jan 23. PMID 29338466